CLINICAL TRIAL: NCT03405571
Title: A Prospective Validation of the 4TS Risk Assessment Model in the Prevention of Venous Thromboembolism in Patients With Plasma Cell Dyscrasias. ROADMAP-MM
Brief Title: Validation of the 4TS RAM in the Prevention of Venous Thromboembolism in Patients With Plasma Cell Dyscrasias.
Acronym: ROADMAP-MM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Collaborators: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Meletios A. Dimopoulos, Professor MA Dimopoulos, University of Athens
Other Study IDs: ROADMAP-MM
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma; Venous Thromboembolism
MeSH Terms: conditions — Multiple Myeloma; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Patients with newly diagnosed symptomatic multiple myeloma per IMWG criteria prior to therapy initiation are enrolled in the study. The aim of the study is to investigate clinical and disease related risk factors for venous thromboembolism (VTE) in these patients as well as possible biomarkers of hypercoagulability linked with the occurrence of venous thromboembolism at diagnosis and during the disease course. The purpose is to create a risk assessment model for VTE in newly diagnosed multiple myeloma patients and make the model more accurate by combining relevant clinical and disease characteristics with biomarkers of cellular and plasma hypercoagulability. A standardized clinical research form is completed for all patients at baseline, 3, 6 and 12 month follow up to include relevant clinical, patient-related, disease-related and treatment related data. Blood sampling also takes place at baseline and 3,6,12 months to assess multiple biomarkers of plasma and cellular hypercoagulability. In addition lowe limb ultrasound is performed at baseline, 6 and 12 months. The primary endpoint is VTE occurrence. Following the elaboration of the ROADMAP-CAT-MM risk assessment model we will prospectively validate it. We expect that patients who are classified, as high risk according to the ROADMAP-CAT-MM will experience symptomatic VTE more frequently and will have higher morbidity and mortality rates during the follow-up. The prospective validation of the ROADMAP-CAT-MM will provide guidance for the use and choice of thromboprophylaxis in these patients and will identify high risk patients eligible for thromboprophylaxis with low molecular weight heparin (tinzaparin).

In addition to symptomatic patients with multiple myeloma the study aims to investigate VTE risk in all plasma cell dyscrasias and will recruit patients with monoclonal gammopathy of undetermined significance, asymptomatic multiple myeloma, primary amyloidosis and Waldenström's macroglobulinemia.

DETAILED DESCRIPTION:
Hypothesis: We expect that patients who are classified, as high risk according to the ROADMAP-CAT-MM will experience symptomatic VTE more frequently and will have higher morbidity and mortality rates during the follow-up. The prospective validation of the ROADMAP-CAT-MM (combined or not with biomarkers of hypercoagulability) will allow to identify patients eligible for long-term thromboprophylaxis with intermediate dose of tinzaparin.

Objectives of the study Primary objective: using the ROADMAP-CAT-MM we will identify high risk patients who will be eligible for long-term thromboprophylaxis.

Secondary objective: to identify patients with biological resistance to the fixed dose of postoperative thromboprophylaxis LMWH and to evaluate its clinical relevance.

End-points of the study Primary end-point: the occurrence of symptomatic VTE (DVT and/or PE) and asymptomatic DVT, or superficial venous thrombosis of the lower or upper limb, central vein catheter thrombosis or venous thrombosis of rare localization. Venous thrombosis has to be confirmed with any of the following assays: echo-Doppler, CT or MRI angiography, or scintigraphy or CT scan. Occurrence of asymptomatic venous thrombosis found during routine imaging for staging will also be included in the primary end point. Combined end-point including all the above types of venous thrombosis will also be evaluated.

Secondary end-points: mortality, major bleeding, cancer evolution and morbidity during follow-up.

Study design: The proposed project is a prospective observational event driven study. The cohort of multiple myeloma patients will be composed by pre-specified groups (1)Group MM-ASA : patients with plasma cell dyscrasias on treatment with aspirin (2) Group MM-LMWH: patients with plasma cell dyscrasias on treatment with usual prophylactic doses of tinzaparin (3) Group MM-No: patients with plasma cell dyscrasias not receiving any antithrombotic treatment Inclusion criteria: Patients with diagnosis of active multiple myeloma, asymptomatic multiple myeloma, Patients with MGUS, Patients with amyloidosis, Patients with Waldenström's macroglobulinemia, A detailed data base on clinical profile of the patients (stage, previous treatments, etc) and the presence of VTE risk factors will be constructed.

Procedures Clinical assessment and follow up: Clinical data will be recorded in pre-specified CRF: At the inclusion, at 3, 6 and 12 months patient records will be checked.

Assessment of biomarkers of cellular and plasma hypercoagulability Blood samples: At the routine follow up and according to the established practice of the clinical investigation centers and the standardized institutional practice for laboratory monitoring of the patients, blood samples will be obtained after atraumatic vein puncture according to standardized procedure, in order to assess biomarkers of hypercoagulability. No additional blood samples to those routinely taken, will be required. The tests required for the present study will be performed using the residual blood from that required for routine laboratory tests.

Blood will be collected in 2 Vacutainer tubes (5 ml tubes, containing 0.109 mol/L trisodium citrate - 1 volume trisodium citrate to 9 volumes blood). Antecubital vein puncture will be performed using 21G needles, or blood will be withdrawn from a recently (within 2-3 minutes) placed peripheral venous cathether (20G). Following a double centrifugation at 1500 x g for 20 minutes, platelet-poor plasma (PPP) will be prepared within 30 minutes after vein puncture. Plasma will be stored in -80 degrees. Blood samples will be collected at the baseline visit and after 3, 6, and 12 months.

Laboratory assays Platelet activation markers: Flow cytometry : platelet derived microparticles expressing P-Selectin Blood coagulation assays: Thrombin generation in platelet poor and platelet rich plasma (Thrombinoscope assay), PPL-Clotting time Other tests, Fibrinogen, D-Dimers Systematic compression ultrasound examination of external iliac and lower extremity veins: A systematic compression ultrasound examination will be performed by one operator, unaware of the history and treatment assignments, at the following time-points: baseline, at 6 months, at 1 year/ end of the study and at the event. All compression ultrasound examinations will be digitally recorded for further adjudication if needed. Statistics A power calculation is difficult to make because this study concerns a pilot study. The results of the tests will be compared using the Student t-test or a non-parametric test where appropriate.

Ethical consideration: The study will be conducted according to the principles of the last Declaration of Helsinki and in accordance with the Medical Research Involving Human Subjects Act (WMO) and other regulations, guidelines and acts.

Patients recruitment, benefits and risks: Screening and informed consent will be taken by the investigator or the Clinical Research Assistant (CRA). The investigator will be responsible for blood collection. Plasma samples will be prepared and stored at the investigation center under the responsibility of the Investigator. The CRA will visit the Centers weakly, will collect the CRF and will confirm the good quality of the plasma samples. The CRA will be responsible for the follow up of the patients (the telephone interview and files revision). The CRA will centralize the samples at the Institut on Thrombosis and Haemostasis and will be responsible for the expedition to the Core Lab in Paris.The CRA will construct the combined data base of clinical and laboratory data.

No benefits can be expected for individual patients who participate in this study. However, more information on this subject can help in the identification of patients with the highest risk of venous thrombosis. These patients might in the future benefit from prophylactic anticoagulants. If knowledge on this subject becomes incorporated into patient care, it will be in the same group of patients who participate in the present study. Results from this study, i.e. microparticle activity, will not have an influence on regular patient care, because of its experimental character. Patients can refuse to participate in the study for any reason, without consequences for regular treatment. Also, the investigator can decide to withdraw a subject from the study for medical reasons. Risks are not to be expected, because of the observational character of this study. The burden of the study is low, because it only includes a single blood withdrawal. Each patient has to make his or her own comparative assessment and decide on a voluntary base. The Medical Ethical Committee has given us dispensation from the obligation to provide insurance.

ADMINISTRATIVE ASPECTS: All investigators will have access to the research data in a coded form. Patient data will be coded and the code will be stored and taken care of by the responsible investigator. Patient material will be stored in a coded form.

ELIGIBILITY:
Inclusion Criteria:

* Newly Diagnosed patients with symptomatic multiple myeloma
* Previously untreated patients

Exclusion Criteria:

* Age younger than 18 years
* Life expectancy less than 6 months
* Ongoing pregnancy, major psychiatric disorders
* Recent (<6 months) episode of VTE or acute coronary syndrome
* Active anticoagulant treatment (for any indication)
* Scheduled open elective curative surgery under general anesthesia for abdominal or pelvic or lung cancer last 3 months
* Hospitalization due to stroke or acute coronary syndrome or congestive heart failure or acute respiratory failure the last 3 months
* Eligible patients had not undergone any surgery in the preceding 3 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed, treatment naïve patients with MM recruited from the outpatient Hematology and Oncology Unit of the Clinical Therapeutics Department (Alexandra Hospital, Athens, Greece)
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Symptomatic venous thromboembolism | 12 months
  Symptomatic objectively confirmed venous thromboembolism

SECONDARY OUTCOMES:
Mortality | 12 months
  deaths per 1000 persons per year
Major Bleeding | 12 months
  major bleeding event
Disease progression | 12 months
  Progressive disease based on the international myeloma working group criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandra Hospital , Department of Clinical Therapeutics, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No